CLINICAL TRIAL: NCT06765759
Title: Impact of Prone Position Duration and Sex Differences on Ventilation and Oxygenation in COVID-19 ARDS Patients: a Retrospective Cohort Study.
Brief Title: Prone Duration in COVID-19 ARDS
Acronym: PRODUR-CARDS
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Oguzhan Kayhan, Lecturer, Istanbul University - Cerrahpasa
Other Study IDs: 2023/789
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: COVID - 19; Acute Respiratory Distress Syndrome (ARDS)
Keywords: COVID - 19; Acute Respiratory Distress Syndrome; Prone Position; Sex
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Short Prone: The group of patients who remained in prone position for 16-24 hours
- Long Prone: The group of patients who remained in prone position for 24-36 hours

SUMMARY:
The aim of this observational study is to learn the effects of prone position duration on patient outcomes in patients with severe acute respiratory distress syndrome (ARDS) due to Coronavirus Disease - 2019 (COVID-19). The main question it aims to answer is:

Does the length of prone position duration affect gas exchange in patients with severe ARDS and is there a difference between genders in this regard? The differences in gas exchange between those who have been in prone position for 16-24 hours and those who have been in prone position for 24-36 hours as part of severe ARDS treatment will be examined.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* hospitalized for more than 48 hours
* patients diagnosed with COVID-19
* intubated patients
* underwent prone positioning for longer than 16 hours starting from the first session

Exclusion Criteria:

* Pregnant females
* Patients under the age of 18
* Those who did not reach 16 hours duration of prone position for various reasons (unintentional extubation, ventilation problems, hemodynamic instability, cardiac arrest-prearrest)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of Covid-19 ARDS patients hospitalized in the tertiary intensive care unit of a university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Calculation of PaO2/FiO2 ratio during short and long prone periods | At each prone session, calculation will be started one hour before the pronation and finished one hour after returning supine.
  Partial arterial oxygen pressure/Fraction of inspired oxygen (PaO2/FiO2) ratio changes before, during and after pronation at each group will be calculated.

SECONDARY OUTCOMES:
Measurement of PaCO2 during short and long prone periods | At each prone session, measurement will be started one hour before the pronation and finished one hour after returning supine.
  Partial arterial carbon dioxide pressure (PaCO2) changes before, during and after pronation at each group will be measured.
Measurement of PEEP during short and long prone periods | At each prone session, measurement will be started one hour before the pronation and finished one hour after returning supine.
  Positive end-expiratory pressure (PEEP) changes before, during and after pronation at each group will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University - Cerrahpaşa, Cerrahpaşa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Approval was not obtained from the institute's ethics committee for sharing patient data with an international registry.